CLINICAL TRIAL: NCT01332175
Title: The Effects of Provent® on Obstructive Sleep Apnea During Continuous Positive Airway Pressure Therapy Withdrawal: a Randomised Controlled Trial.
Brief Title: The Effects of Provent® on Obstructive Sleep Apnea During Continuous Positive Airway Pressure Therapy Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK-1600
Record Dates: First submitted 2011-04-01; First posted 2011-04-08 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Provent (Active Comparator)
  Interventions: Device: Provent®
- Placebo-Provent (Placebo Comparator)
  Interventions: Device: Provent®; Device: Placebo-Provent®
- CPAP (Active Comparator)
  Interventions: Device: Provent®; Procedure: CPAP

INTERVENTIONS:
Device: Provent® — Nightly use of Provent® versus Placebo-Provent® versus CPAP
Device: Placebo-Provent® — Nightly use of Provent® versus Placebo-Provent® versus CPAP
  Arms: Placebo-Provent
Procedure: CPAP — Nightly use of Provent® versus Placebo-Provent® versus CPAP
  Arms: CPAP

SUMMARY:
Randomised, placebo-controlled trial of continuous positive airway pressure therapy (CPAP) versus Provent® and Placebo-Provent® to define the effects of Provent® on the severity of obstructive sleep apnea, daytime symptoms as well as on measures of cardiovascular risk.

DETAILED DESCRIPTION:
Randomised, placebo-controlled trial of Provent® versus Placebo-Provent® versus continuous positive airway pressure therapy (CPAP) to define the effects of Provent® on the severity of obstructive sleep apnea, daytime symptoms as well as on measures of cardiovascular risk in patients with obstructive sleep apnea.

Patients successfully treated with CPAP will be randomised to one of three arms for a duration of 2 weeks:

1. Withdraw CPAP and use Provent®
2. Withdraw CPAP and use Placebo-Provent®
3. Continue treatment with CPAP

ELIGIBILITY:
Inclusion criteria:

1. Objectively confirmed obstructive sleep apnoea (at the time of original diagnosis) with an oxygen desaturation index (ODI, >4% dips) of between 10 and 50/h and an ESS of >10 (these thresholds will exclude subjects with borderline and very severe forms of OSA in whom there may be a disproportionate treatment effect).
2. Currently >10/h oxygen desaturations (>4% dips) during an ambulatory nocturnal pulse oximetry performed at the end of a 4-night period without CPAP.
3. Treated with NCPAP for more than 12 months, minimum compliance 4h per night.
4. Current ESS < 10.
5. Written informed consent.

Exclusion criteria:

1. Previous ventilatory failure (awake resting arterial oxygen saturation <93% or arterial PCO2 > 6kPa).
2. Unstable, untreated coronary or peripheral artery disease, severe arterial hypertension (>180/110mmHg).
3. Previously diagnosed with Cheyne-Stokes breathing.
4. Current professional driver.
5. Any sleep related accident.
6. Age <20 or >75 years at trial entry.
7. History of chronic nasal obstruction.
8. Mental or physical disability precluding informed consent or compliance with the protocol .
9. Non-feasible trial follow-up (for example, distance from follow-up centre, physical inability).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sleep apnoea severity, daytime symptoms of sleep apnoea | 2 weeks

SECONDARY OUTCOMES:
Blood pressure | 2 weeks
  Comparison of changes in systolic and diastolic blood pressure from baseline to follow-up at 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Leading Physician, Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (3):
- Switzerland (2):
  - Cantonal Hospital Munsterlingen, Departement of Internal Medicine, Pulmonary Division, Münsterlingen
  - University Hospital Zurich, Pulmonary Division, Zurich
- Churchill Hospital, Oxford Centre for Respiratory Medicine, Oxford, United Kingdom

REFERENCES:
- [Derived] Crook S, Sievi NA, Bloch KE, Stradling JR, Frei A, Puhan MA, Kohler M. Minimum important difference of the Epworth Sleepiness Scale in obstructive sleep apnoea: estimation from three randomised controlled trials. Thorax. 2019 Apr;74(4):390-396. doi: 10.1136/thoraxjnl-2018-211959. Epub 2018 Aug 12. PMID 30100576
- [Derived] Stoberl AS, Schwarz EI, Haile SR, Turnbull CD, Rossi VA, Stradling JR, Kohler M. Night-to-night variability of obstructive sleep apnea. J Sleep Res. 2017 Dec;26(6):782-788. doi: 10.1111/jsr.12558. Epub 2017 May 26. PMID 28548301
- [Derived] Schwarz EI, Schlatzer C, Rossi VA, Stradling JR, Kohler M. Effect of CPAP Withdrawal on BP in OSA: Data from Three Randomized Controlled Trials. Chest. 2016 Dec;150(6):1202-1210. doi: 10.1016/j.chest.2016.07.012. Epub 2016 Jul 21. PMID 27452767
- [Derived] Rossi VA, Winter B, Rahman NM, Yu LM, Fallon J, Clarenbach CF, Bloch KE, Stradling JR, Kohler M. The effects of Provent on moderate to severe obstructive sleep apnoea during continuous positive airway pressure therapy withdrawal: a randomised controlled trial. Thorax. 2013 Sep;68(9):854-9. doi: 10.1136/thoraxjnl-2013-203508. Epub 2013 May 30. PMID 23723343